CLINICAL TRIAL: NCT02109354
Title: Phase 1b Randomized Double Blind Placebo Controlled Clinical Trial to Evaluate the Safety and Immunogenicity of the Vaccine Regimen ALVAC-HIV (vCP1521) Followed by AIDSVAX® B/E in Healthy, HIV-1 Uninfected Adult Participants in South Africa
Brief Title: Safety of and Immune Response to Vaccination With 2 Experimental HIV Vaccines in Healthy Adults
Acronym: HVTN 097
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HIV Vaccine Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 097
Record Dates: First submitted 2013-12-12; First posted 2014-04-09 (Estimated); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: HIV Infection
Keywords: HIV infection; Vaccine
MeSH Terms: conditions — HIV Infections | interventions — AIDSVAX; AIDSVAX B-E; HIV Envelope Protein gp120; Hepatitis B Vaccines; Engerix-B; Tetanus Toxoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HIV Regimen + Tetanus and HBV Vaccines (Active Comparator): Participants will receive a tetanus vaccine injection (tetanus toxoid vaccine), followed by 2 injection of an experimental canarypox HIV vaccine (ALVAC-HIV; months 1, 2), than 2 injection of a protein HIV vaccine boost (AIDSVAX B/E; months 4, 7), followed by a hepatitis B vaccine series (months 7.5, 8.5, 13)
  Interventions: Biological: ALVAC-HIV; Biological: AIDSVAX B/E; Biological: Hepatitis B vaccine; Biological: Tetanus toxoid vaccine
- HIV Vaccine Regimen (Active Comparator): Participants will receive a placebo for tetanus vaccine by injection (placebo tetanus toxoid vaccine), followed by 2 injection of an experimental canarypox HIV vaccine (ALVAC-HIV; months 1, 2), than 2 injection of a protein HIV vaccine boost (AIDSVAX B/E; months 4, 7), followed by a placebo for hepatitis B vaccine series (months 7.5, 8.5, 13)
  Interventions: Biological: ALVAC-HIV; Biological: AIDSVAX B/E; Biological: Placebo for hepatitis B vaccine; Biological: Placebo for tetanus vaccine
- Tetanus and HBV Vaccines (Placebo Comparator): Participants will receive a tetanus vaccine injection (tetanus toxoid vaccine), followed by 2 injection of a placebo for the experimental canarypox HIV vaccine (placebo for ALVAC-HIV; months 1, 2), than 2 injection of a placebo protein HIV vaccine boost (placebo for AIDSVAX B/E; months 4, 7), followed by a hepatitis B vaccine series (months 7.5, 8.5, 13)
  Interventions: Biological: Placebo for ALVAC-HIV; Biological: Placebo for AIDSVAX B/E; Biological: Hepatitis B vaccine; Biological: Tetanus toxoid vaccine

INTERVENTIONS:
Biological: ALVAC-HIV — Formulated as a lyophilized vaccine for injection and is reconstituted with 1.05 mL of sterile Sodium Chloride solution (0.4% NaCl) for a single 1 mL dose of >1.0 x 106 CCID50/mL, to administer intramuscularly (IM).
  Other Names: vCP1521
  Arms: HIV Regimen + Tetanus and HBV Vaccines; HIV Vaccine Regimen
Biological: AIDSVAX B/E — 300 mcg of subtype B (MN) HIV gp120 glycoprotein and 300 mcg of subtype E (A244) HIV gp120 glycoprotein adsorbed onto 600 mcg of aluminum hydroxide gel adjuvant. Each vial contains 1.2 mL of sterile suspension, to administer 1 mL IM.
  Other Names: gp120
  Arms: HIV Regimen + Tetanus and HBV Vaccines; HIV Vaccine Regimen
Biological: Placebo for ALVAC-HIV — A sterile, lyophilized product that consists of a mixture of virus stabilizer, and freeze drying medium and is reconstituted with 1.05 mL of sterile Sodium Chloride (0.4% NaCl) for a single 1 mL dose, to administer IM.
  Arms: Tetanus and HBV Vaccines
Biological: Placebo for AIDSVAX B/E — Sodium Chloride for Injection, 0.9% administered IM.
  Arms: Tetanus and HBV Vaccines
Biological: Hepatitis B vaccine — Each 1 mL dose contains 20 mcg of hepatitis B surface antigen (HBsAg) adsorbed onto 500 mcg aluminum as aluminum hydroxide, to administer IM.
  Other Names: HBV vaccine; ENGERIX-B
  Arms: HIV Regimen + Tetanus and HBV Vaccines; Tetanus and HBV Vaccines
Biological: Tetanus toxoid vaccine — The active ingredient is tetanus toxoid (≥ 40 I.U. / 0.5 mL) adsorbed on aluminium hydroxide dihydrate (600 mcg of aluminium), to administer IM.
  Other Names: Tetanus vaccine; Tetavax
  Arms: HIV Regimen + Tetanus and HBV Vaccines; Tetanus and HBV Vaccines
Biological: Placebo for hepatitis B vaccine — Sodium Chloride for Injection, 0.9% administered IM.
  Arms: HIV Vaccine Regimen
Biological: Placebo for tetanus vaccine — Sodium Chloride for Injection, 0.9% administered IM.
  Arms: HIV Vaccine Regimen

SUMMARY:
The HIV Vaccine Trials Network (HVTN) is doing a study to test 2 experimental HIV vaccines in combination with 2 licensed vaccines for tetanus and hepatitis B. HIV is the virus that causes AIDS. Tetanus is an infection that causes muscular spasms. Hepatitis B is a virus that can cause liver failure.

About 100 people will take part in this study at multiple sites. The US National Institutes of Health (NIH) is paying for the study.

We are doing this study to answer several questions.

* Are the HIV study vaccines safe to give to people?
* Are people able to take the HIV study vaccines without becoming too uncomfortable?
* How do people's immune systems respond to the HIV study vaccines? (Your immune system protects you from disease.)
* Can people's immune responses to a tetanus or hepatitis B vaccines help us understand how their immune systems might respond to the HIV study vaccines?
* Is there a common immune response to licensed vaccines like the tetanus and hepatitis B vaccines?

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 40 years
* Access to a participating HVTN CRS and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: volunteer demonstrates understanding of this study; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Agrees not to enroll in another study of an investigational research agent
* Good general health as shown by medical history, physical exam, and screening laboratory tests
* Willingness to receive tetanus and Hepatitis B vaccination
* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks, amenable to HIV risk reduction counseling, and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit
* Assessed by the clinic staff as being at "low risk" for HIV infection
* Hemoglobin ≥ 11.0 g/dL for volunteers who were born female, ≥ 13.0 g/dL for volunteers who were born male
* White blood cell count = 3,300 to 12,000 cells/mm3
* Total lymphocyte count ≥ 800 cells/mm3
* Remaining differential either within institutional normal range or with site physician approval
* Platelets = 125,000 to 550,000/mm3
* Chemistry panel: alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase < 1.25 times the institutional upper limit of normal; creatinine ≤ institutional upper limit of normal.
* Negative HIV-1 and -2 blood test: Sites may use locally available assays that have been approved by HVTN Laboratory Operations.
* Negative Hepatitis B surface antigen (HBsAg)
* Negative Hepatitis B core antibody (HBcAb)
* Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive
* Normal urine:

  * Negative urine glucose,
  * Negative or trace urine protein, and
  * Urinalysis (dipstick) for blood no greater than 1+ (if trace or 1+ hemoglobin is present on dipstick, a microscopic urinalysis with red blood cells levels within institutional normal range).
* Volunteers who were born female: negative serum or urine β human chorionic gonadotropin (β-HCG) pregnancy test performed prior to vaccination on the day of initial vaccination
* Reproductive status: A volunteer who was born female must:

  * Agree to consistently use effective contraception (see Appendix C) for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit. Effective contraception for participants in South Africa is defined as using 2 methods, including the following:

    * Condoms (male or female) with or without a spermicide,
    * Diaphragm or cervical cap with spermicide,

PLUS 1 of the following methods:

* Intrauterine device (IUD),
* Hormonal contraception (in accordance with South African contraception guidelines), or

  * Successful vasectomy in the male partner (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy);
  * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation;
  * Or be sexually abstinent.

    * Volunteers who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Exclusion Criteria:

* Blood products received within 120 days before first vaccination
* Investigational research agents received within 30 days before first vaccination
* Body mass index (BMI) ≥ 40; or BMI ≥ 35 with 2 or more of the following: age > 45, systolic blood pressure > 140 mm Hg, diastolic blood pressure > 90 mm Hg, current smoker, known hyperlipidemia
* Intent to participate in another study of an investigational research agent during the planned duration of the HVTN 097 study
* Pregnant, breastfeeding or lactating
* History of Hepatitis B viral infection
* History of tetanus disease Vaccines and other Injections
* HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 097 PSRT will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial. Exceptions may be made for vaccines that have subsequently undergone licensure by the South Africa Medicines Control Council (MCC). For volunteers who have received control/placebo in an experimental vaccine trial, the HVTN 097 PSRT will determine eligibility on a case-by-case basis. For volunteers who have received an experimental vaccine(s) greater than 5 years ago, eligibility for enrollment will be determined by the HVTN 097 PSRT on a case-by-case basis.
* Live attenuated vaccines other than influenza vaccine received within 30 days before first vaccination or scheduled within 14 days after injection (eg, measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Influenza vaccine or any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (eg, pneumococcal, Hepatitis A)
* Any requirement to receive an HBV vaccine other than the HBV vaccine given during the study period.
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination
* Known to have received a tetanus vaccination within the last 5 years prior to first vaccination.
* Immunosuppressive medications received within 168 days before first vaccination. (Not excluded: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatitis; or [4] a single course of oral/parenteral corticosteroids at doses < 2 mg/kg/day and length of therapy < 11 days with completion at least 30 days prior to enrollment.
* Serious adverse reactions to vaccines including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded: a volunteer who had a nonanaphylactic adverse reaction to pertussis vaccine as a child.)
* History of allergic reaction to yeast
* History of allergic reaction to HBV or tetanus vaccine or any component of the vaccines or placebo, including eggs, egg products, or neomycin
* Immunoglobulin received within 60 days before first vaccination
* Autoimmune disease
* Immunodeficiency
* Untreated or incompletely treated syphilis infection
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response,
  * A process that would require medication that affects the immune response,
  * Any contraindication to repeated injections or blood draws,
  * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
  * A condition or process for which signs or symptoms could be confused with reactions to vaccine, or
  * Any condition specifically listed among the exclusion criteria below.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-TB prophylaxis or therapy
* Asthma other than mild or moderate, well-controlled asthma. (Symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program (NAEPP) Expert Panel report).

Exclude a volunteer who:

* Uses a short-acting rescue inhaler (typically a β 2 agonist) daily, or
* Uses high dose inhaled corticosteroids, or
* In the past year has either of the following:

  * Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids;
  * Needed emergency care, urgent care, hospitalization, or intubation for asthma.

    * Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes.)
    * Thyroidectomy, or thyroid disease requiring medication during the last 12 months
    * Hypertension:
* If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently ≤ 140 mm Hg systolic and ≤ 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be ≤ 150 mm Hg systolic and ≤ 100 mm Hg diastolic. For these volunteers, blood pressure must be ≤ 140 mm Hg systolic and ≤ 90 mm Hg diastolic at enrollment.
* If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure ≥ 150 mm Hg at enrollment or diastolic blood pressure ≥ 100 mm Hg at enrollment.

  * Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
  * Malignancy (Not excluded: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure. or who is unlikely to experience recurrence of malignancy during the period of the study)
  * Seizure disorder: History of seizure(s) within past three years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
  * Asplenia: any condition resulting in the absence of a functional spleen
  * History of hereditary angioedema, acquired angioedema, or idiopathic angioedema.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2013-06-18 (Actual); Primary Completion 2015-02-02 (Actual); Study Completion 2015-02-02 (Actual)

PRIMARY OUTCOMES:
Frequency of local and systemic reactogenicity signs and symptoms, laboratory measures of safety, and a line listing of all AEs meeting DAIDS criteria for expedited reporting. | 13.5 months
HIV-specific total IgG and IgA binding antibody responses as assessed by multiplex assay | 2 weeks following the final vaccination of ALVAC-HIV + AIDSVAX B/E.
Neutralizing antibody magnitude and breadth against tier 1 and tier 2 HIV-1 isolates as assessed by area under the magnitude-breadth curves | 2 weeks following the final vaccination of ALVAC-HIV + AIDSVAX B/E.
Magnitude and frequency of HIV-specific CD4+ and CD8+ T-cell responses as assessed by flow cytometry at 2 weeks following the final vaccination of ALVACHIV + AIDSVAX B/E. | 2 weeks post final vaccination of ALVACHIV + AIDSVAX B/E
Frequency of severe local and systemic reactogenicity signs and symptoms (pain, tenderness, erythema, induration, fever, malaise/fatigue, myalgia, headache, nausea, vomiting, chills, arthralgia) | 3 days after each vaccine dose
Frequency of AEs by body system, Medical Dictionary for Regulatory Activities (MedDRA) preferred term, severity, and assessed relationship to study products | 30 days after each vaccine dose
Frequency of SAEs, adverse events of special interest (AESIs; Appendix K), and new chronic conditions (requiring medical intervention for ≥ 30 days) throughout the study | 19.5 months
Composite of safety laboratory measures: white blood cells, neutrophils, lymphocytes, hemoglobin, platelets, alanine aminotransferase, aspartate aminotransferase, alkaline phosphate, and creatinine at baseline and following vaccinations | 19.5 months
Frequency of AEs leading to early participant withdrawal or early discontinuation of study products administration throughout the study. | 19.5 months
Occurrence and level of vaccine-induced IgG binding Ab to gp120 and V1V2 scaffold | 2 week sand 6 months post first-boost

SECONDARY OUTCOMES:
Anti-V1/V2 IgG binding antibody responses as assessed by multiplex assay | 2 weeks following the final vaccination of ALVAC-HIV + AIDSVAX B/E
Titers of antibody-dependent cellular cytotoxicity (ADCC) or antibody-dependent cellular viral inhibition (ADCVI)-mediating antibodies | 2 weeks following the final vaccination of ALVAC-HIV + AIDSVAX B/E.
HIV-specific IgG subclass (IgG1-IgG4) characterization as determined by HIV-1 multiplex Ab assay | 2 weeks following the final vaccination of ALVAC-HIV + AIDSVAX B/E.
Avidity indices for Env-specific antibodies | 2 weeks following the final vaccination of ALVAC-HIV + AIDSVAX B/E.
HIV-capturing non-neutralizing antibodies as assessed by competitive virus capture assay | 2 weeks following the final vaccination of ALVAC-HIV + AIDSVAX B/E.
B-cell ELISpot to quantify Env-specific antibody-producing B cells | 2 weeks following the final vaccination of ALVAC-HIV + AIDSVAX B/E.
Expression of cytokines (eg, IL-10, IL-13) by multiplex bead array following antigen-specific stimulation of peripheral blood mononuclear cells (PBMC) | 2 weeks following the final vaccination of ALVAC-HIV + AIDSVAX B/E.
Changes in PBMC gene expression relative to prevaccine levels of key genes expected to change. | 19.5 months
Concentrations of cytokines and chemokines in serum and/or plasma samples. | 19.5 months
Cell phenotype assessed by flow cytometric analysis of PBMC subsets. | 19.5 months
HIV-specific humoral and cellular responses 6 months following the final vaccination of ALVAC-HIV + AIDSVAX B/E. | 6 months following the final vaccination of ALVAC-HIV + AIDSVAX B/E.
HIV-specific humoral and cellular responses 2 weeks following the final vaccination of ALVAC-HIV + AIDSVAX B/E. | 2 weeks following the final vaccination of ALVAC-HIV + AIDSVAX B/E.
Occurrence and level of vaccine-induced IgG binding Ab to gp120 and V1V2 scaffold | 2 weeks and 6 months post second-boost as assessed by multiplex assay
Occurrence, magnitude, character and breadth of systemic HIV-specific binding antibody responses as assessed by multiplex assay | baseline (Time 0 prior to first boost), at 2 weeks and at 6 months following each boost, and at 12 months following the first boost including subtype, subclass and IgG binding Ab to V3 epitopes
HIV-specific systemic CD4+ and CD8+ T-cell responses | baseline (Time 0 prior to first boost), at 2 weeks and at 6 months following each boost, and at 12 months following the first boost
Systemic neutralizing antibody magnitude and breadth against tier 1 and, if applicable, tier 2 HIV-1 isolates as assessed by area under the magnitude-breadth curves | 2 weeks following each boost
Functional humoral immune responses including ADCC and HIV virus capture | 19.5 months
Additional immunogenicity assays may be performed on blood and mucosal samples, including on samples from other timepoints, based on the HVTN Laboratory Assay Algorithm. | 19.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Gray, MD, Study Chair — Perinatal HIV Research Unit
Locations (3):
- South Africa (3):
  - Emavundleni Desmond Tutu HIV Centre CRS, Cape Town, Western Cape
  - Aurum Institute for Health Research, Klerksdorp
  - Perinatal HIV Research Unit, Soweto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moodie Z, Li SS, Giorgi EE, Williams LD, Dintwe O, Carpp LN, Chen S, Seaton KE, Sawant SS, Zhang L, Heptinstall J, Liu S, Grunenberg N, Tomaka F, Rerks-Ngarm S, Pitisuttithum P, Nitayaphan S, Ake JA, Vasan S, Pantaleo G, Frank I, Baden LR, Goepfert PA, Keefer M, Chirenje M, Hosseinipour MC, Mngadi K, Laher F, Garrett N, Bekker LG, De Rosa S, Andersen-Nissen E, Kublin JG, Lu S, Gilbert PB, Gray GE, Corey L, McElrath MJ, Tomaras GD. A polyvalent DNA prime with matched polyvalent protein/GLA-SE boost regimen elicited the most robust and broad IgG and IgG3 V1V2 binding antibody and CD4+ T cell responses among 13 HIV vaccine trials. Emerg Microbes Infect. 2025 Dec;14(1):2485317. doi: 10.1080/22221751.2025.2485317. Epub 2025 Apr 7. PMID 40190112
- [Derived] Zhao LP, Fiore-Gartland A, Carpp LN, Cohen KW, Rouphael N, Fleurs L, Dintwe O, Zhao M, Moodie Z, Fong Y, Garrett N, Huang Y, Innes C, Janes HE, Lazarus E, Michael NL, Nitayaphan S, Pitisuttithum P, Rerks-Ngarm S, Robb ML, De Rosa SC, Corey L, Gray GE, Seaton KE, Yates NL, McElrath MJ, Frahm N, Tomaras GD, Gilbert PB. Landscapes of binding antibody and T-cell responses to pox-protein HIV vaccines in Thais and South Africans. PLoS One. 2020 Jan 30;15(1):e0226803. doi: 10.1371/journal.pone.0226803. eCollection 2020. PMID 31999736
- [Derived] Lazarus EM, Otwombe K, Adonis T, Sebastian E, Gray G, Grunenberg N, Roux S, Churchyard G, Innes C, Laher F. Uptake of genital mucosal sampling in HVTN 097, a phase 1b HIV vaccine trial in South Africa. PLoS One. 2014 Nov 17;9(11):e112303. doi: 10.1371/journal.pone.0112303. eCollection 2014. PMID 25401780